CLINICAL TRIAL: NCT05542667
Title: Comparative Evaluation of Giomer Varnish vs Fluoride Varnish as Desensitizing Agents Among a Group of Children With Molar Incisor Hypomineralization : A Controlled Clinical Trial
Brief Title: Comparative Evaluation of Giomer Varnish vs Fluoride Varnish as Desensitizing Agents in Teeth With MIH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ethar khaled hassan ahmed swidan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8484
Record Dates: First submitted 2022-08-17; First posted 2022-09-15 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Giomer varnish (Active Comparator): PRG coat barrier by SHOFU is varnish based on a new technology named Giomer by incorporating pre-reacted glass ionomer particles, so varnish contains GI particles embedded in a resin matrix, it should be applied once per year since it is the only varnish in the market that is light cured so it is more durable than others.
  Interventions: Combination Product: Giomer varnish
- Fluoroide varnish (Active Comparator): Bifluorid 10 by VOCO is a varnish containing 5% sodium fluoride and 5 % calcium fluoride, it should be applied once each 6 months by a professional dentist and it tends to decrease the hypersensitivity of the teeth as well as decrease the risk of caries.
  Interventions: Combination Product: Fluoride varnish

INTERVENTIONS:
Combination Product: Giomer varnish — * After dryness and isolation are accomplished, Giomer varnish ( PRG coat barrier, by Shofu) will be applied once at the first treatment visit, one drop of PRG Coat Barrier ACTIVE will be added to the container provided in the package containing PRG Coat Barrier BASE the materials will be mixed together with a disposable tip provided by the kit a thin layer is to be applied and left untouched for 3 seconds according to manufacturer instructions and finally varnish is to be light-cured.
  Arms: Giomer varnish
Combination Product: Fluoride varnish — After dryness and isolation are accomplished, fluoride varnish (Biflourid 10, by Voco ) single-use type, the foil in the single-use Bifluorid 10 will be pierced using Micro-Tim brush, then a thin layer of the varnish is to be applied using a micro brush for four sessions at a frequency of one session each week, the varnish will be left undisturbed for 10-20 seconds then air-dried according to manufacturer instructions.
  Arms: Fluoroide varnish

SUMMARY:
this clinical trial's aim is to compare two desensitizing agents available in the market to prove which one is more efficient in children with molar incisor hypomineralization complaining from hypersensitivity

DETAILED DESCRIPTION:
Interventions

The principal investigator will carry out all treatment procedures, and the patients will be assigned.

For both interventions:

1. Informed consent from participating parents.
2. Baseline records photographs and personal data collection .
3. Allocation (concealed by withdrawing a sealed opaque envelope containing eight times folded paper containing the type of desensitizing agent that will be used then writing the patient name and I.D. on it and will be opened in the first visit of treatment).
4. Diagnostic chart with personal, medical, and dental history will be filled.
5. Evaluation of oral health-related quality of life as a baseline, using the Arabic version of the child perception questionnaire-8-10m indicated for children from age 8 to 10 years old, it consists of 25 questions related to oral symptoms (5 questions), functional limitations ( 5 questions), emotional wellbeing (5 questions) and social wellbeing ( 10 questions), responses are made on an ordinal scale ( 0 = never, 1 = once/twice, 2= sometimes, 3= often, 4= every day/ almost every day).
6. Teeth will be cleaned with prophylaxis paste using a low-speed contra brush then teeth will be inspected using a dental mirror and reflected light of the dental unit and the teeth must be moist during the clinical examination to assess the clinical inclusion criteria according to European Academy of Pediatric Dentistry diagnostic criteria.
7. Preoperative, intraoperative, and Postoperative photographs will be taken.
8. Prior to initiation of the treatment, all included teeth will be evaluated for pain in response to an evaporative stimulus using the triple syringe, the air is directed perpendicular to teeth and held at approximately 2 mm for 3 seconds and children are informed to raise their hands or fingers when any discomfort is felt and then the pain is evaluated using the Wong-Baker faces rating scale and Schiff scale.
9. Teeth also are evaluated to thermal stimulus, using an anesthetic carpule refrigerated at 4c for at least 24 hours and the carpule is to be placed in contact with the tooth for 1 to 5 seconds according to child response and pain is to be evaluated as with evaporative stimulus.
10. Application of rubber dam for isolation.
11. Prior to treatment, teeth received prophylaxis using pumice paste, cleaned using the triple water syringe, and dried.

Children will then be allocated into either one of the groups alternatively depending on the desensitizing agent used as follows:

Group I (Experimental group) Giomer varnish. Group II (Control group) Fluoride varnish.

ELIGIBILITY:
Inclusion Criteria:

* Children :

  1. Patients aged between 8 and 10 years old with MIH affected teeth according to European Academy of Pediatric Dentistry diagnostic criteria (Lygidakis et al., 2022)
  2. Systemically healthy.
  3. Cooperative patients who will comply with follow-up visits.
* Teeth:

  1. At least one first molar or one incisor erupted in the oral cavity exhibiting molar incisor hypomineralization.
  2. Teeth representing molar incisor hypomineralization are sensitive.

     -

     Exclusion Criteria:
     * • Children:

  <!-- -->

  1. Undergoing desensitizing treatments in the last 3 months
  2. Occlusal problems such as bruxism.
  3. Cognition problems.
  4. Who used any type of analgesics before treatment.
  5. Undergoing orthodontic treatment.
* Teeth:

  1. Enamel defects as enamel hypoplasia, amelogenesis imperfecta, and dental fluorosis.
  2. Carious teeth.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Absence of pain to the evaporative stimulus | 1 month
  will be measured using wong baker faces rating scale from 0 to 5 , 0 being the better outcome
Absence of pain to the evaporative stimulus | 1 month
  will be measured using schiff scale from 0 to 3 , 0 being the better outcome

SECONDARY OUTCOMES:
Absence of pain to thermal stimulus | 1 month
  will be measured using wong baker faces rating scale from 0 to 5 , 0 being the better outcome
Evaluation of oral health-related quality of life (OHRQoL) | 1 month
  measured using the Arabic child perception questionnaire from age 8-10 years old , contains 25 questions and each answer is rating from 0 to 4 , 0 being the better outcome

IPD SHARING:
Plan to Share IPD: Yes
study protocol ,details about interventions , statistical methods used and results will all be shared with others.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: once the study have been completed